CLINICAL TRIAL: NCT00073424
Title: Cognitive, Behavioral, and Psychosocial Correlates of Medication Adherence in Children and Adolescents With HIV-1 Infection
Brief Title: Factors Affecting Adherence to Anti-HIV Drug Regimens in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: PACTG P1042s; 10107 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2003-11-20; First posted 2003-11-21 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Taking anti-HIV medication consistently and properly is a critical issue for patients with HIV. Drug regimens are complex; when regimens are not taken properly, HIV can become resistant to the drugs. Taking anti-HIV medication properly leads to improved health. Children and adolescents with HIV face unique challenges to taking HIV medication properly. This study will look at the relationship between how children cope with the responsibility for taking medication and the child's language, memory, attention, behavior, and academic skills. This study is open to children and adolescents who are currently enrolled in the PACTG 219C study (Long-Term Effects of HIV Exposure and Infection in Children).

DETAILED DESCRIPTION:
Medication adherence is a critical issue for HIV infected children and adolescents because of drug resistance and the increased complexity of treatment regimens. Children and adolescents with HIV face depression, anxiety, denial, and rebellion that may interfere with their motivation to take medication. Depression and self-perceived social support have been found to predict regimen adherence in adults with HIV. Children with other chronic diseases are less likely to adhere to their medication regimens if they also have behavioral or emotional problems; assessing emotional and behavioral function in children and adolescents with HIV may help in predicting adherence and explaining adherence failure. This study will correlate cognitive, behavioral, and psychosocial functioning with measures of virologic suppression and immunological status, and it will compare self-report and pill count measures of adherence in a randomly selected subset of perinatally infected HIV participants of PACTG 219C.

Children and adolescents currently enrolled in PACTG 219C will be randomly selected for this study, which will last for 48 weeks. At entry, participants will undergo neuropsychological evaluation, including academic achievement, attention, memory, language comprehension, and behavior assessments, and complete a health beliefs questionnaire. Both the participants and their parents or primary caregivers will complete questionnaires at study entry and Weeks 24 and 48. Adherence will be evaluated from self-reported and pill count measures (Weeks 4 and 24) and the PACTG 219C Adherence Module (Weeks 24 and 48).

ELIGIBILITY:
Inclusion Criteria

* HIV-1 perinatal infection
* Already enrolled and in active follow-up in PACTG 219C
* Can communicate in English or Spanish
* On antiretroviral medication regimen at the time of enrollment, regardless of compliance with regimen, with no planned treatment interruptions

Exclusion Criteria

* Acquired HIV via routes other than perinatal transmission or source of HIV infection is unknown
* HIV-2 infection

Ages: 8 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200
Dates: Start 2004-01; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Nichols, PhD, Study Chair — Department of Neurosciences, University of California, San Diego
Locations (36):
- United States (34):
  - UAB, Dept. of Ped., Div. of Infectious Diseases, Birmingham, Alabama
  - Phoenix Children's Hosp., Phoenix, Arizona
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - Usc La Nichd Crs, Los Angeles, California
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - UCSD Mother-Child-Adolescent Program CRS, San Diego, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Univ. of Colorado Denver NICHD CRS, Denver, Colorado
  - Yale Univ. School of Medicine - Dept. of Peds., Div. of Infectious Disease, New Haven, Connecticut
  - Children's National Med. Ctr., ACTU, Washington D.C., District of Columbia
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - South Florida CDTC Ft Lauderdale NICHD CRS, Fort Lauderdale, Florida
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - Med. College of Georgia School of Medicine, Dept. of Peds., Div. of Infectious Diseases, Augusta, Georgia
  - Chicago Children's CRS, Chicago, Illinois
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Univ. of Maryland Med. Ctr., Div. of Ped. Immunology & Rheumatology, Baltimore, Maryland
  - Johns Hopkins Hosp. & Health System - Dept. of Peds., Div. of Infectious Diseases, Baltimore, Maryland
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Springfield, Massachusetts
  - NJ Med. School CRS, Newark, New Jersey
  - SUNY Downstate Med. Ctr., Children's Hosp. at Downstate NICHD CRS, Brooklyn, New York
  - Nyu Ny Nichd Crs, New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - Jacobi Med. Ctr., The Bronx, New York
  - UNC at Chapel Hill School of Medicine - Dept. of Peds., Div. of Immunology & Infectious Diseases, Chapel Hill, North Carolina
  - DUMC Ped. CRS, Durham, North Carolina
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - St. Christopher's Hosp. for Children, Philadelphia, Pennsylvania
  - St. Jude/UTHSC CRS, Memphis, Tennessee
  - Texas Children's Hosp. CRS, Houston, Texas
- Puerto Rico (2):
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan

REFERENCES:
- [Background] Catz SL, Kelly JA, Bogart LM, Benotsch EG, McAuliffe TL. Patterns, correlates, and barriers to medication adherence among persons prescribed new treatments for HIV disease. Health Psychol. 2000 Mar;19(2):124-33. PMID 10762096
- [Background] Gordillo V, del Amo J, Soriano V, Gonzalez-Lahoz J. Sociodemographic and psychological variables influencing adherence to antiretroviral therapy. AIDS. 1999 Sep 10;13(13):1763-9. doi: 10.1097/00002030-199909100-00021. PMID 10509579
- [Background] Rogers AS, Miller S, Murphy DA, Tanney M, Fortune T. The TREAT (Therapeutic Regimens Enhancing Adherence in Teens) program: theory and preliminary results. J Adolesc Health. 2001 Sep;29(3 Suppl):30-8. doi: 10.1016/s1054-139x(01)00289-0. No abstract available. PMID 11530301
- [Background] Gaughan DM, Hughes MD, Oleske JM, Malee K, Gore CA, Nachman S; Pediatric AIDS Clinical Trials Group 219C Team. Psychiatric hospitalizations among children and youths with human immunodeficiency virus infection. Pediatrics. 2004 Jun;113(6):e544-51. doi: 10.1542/peds.113.6.e544. PMID 15173535
- [Result] Farley JJ, Montepiedra G, Storm D, Sirois PA, Malee K, Garvie P, Kammerer B, Naar-King S, Nichols S; PACTG P1042S Team. Assessment of adherence to antiretroviral therapy in perinatally HIV-infected children and youth using self-report measures and pill count. J Dev Behav Pediatr. 2008 Oct;29(5):377-84. doi: 10.1097/DBP.0b013e3181856d22. PMID 18714204
- [Result] Naar-King S, Montepiedra G, Nichols S, Farley J, Garvie PA, Kammerer B, Malee K, Sirois PA, Storm D; PACTG P1042S Team. Allocation of family responsibility for illness management in pediatric HIV. J Pediatr Psychol. 2009 Mar;34(2):187-94. doi: 10.1093/jpepsy/jsn065. Epub 2008 Jun 27. PMID 18586756